CLINICAL TRIAL: NCT04185350
Title: Clinical Evaluation of 68Ga-NOTA-MAL-Cys39-exendin-4 Positron Emission Tomography in the Detection of Insulinoma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, FengWang, Director of Nuclear Medicine, Nanjing First Hospital, Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NJCNMC-GLP-1
Record Dates: First submitted 2019-12-01; First posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Insulinoma
MeSH Terms: conditions — Insulinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-NOTA-MAL-Cys39-exendin-4 PET/CT (Experimental): The patients were injected with 111-185 MBq of 68Ga-NOTA-MAL-Cys39-exendin-4 PET/CT in one dose intravenously and underwent PET/CT scan 60 min later.
  Interventions: Drug: 68Ga-NOTA-MAL-Cys39-exendin-4

INTERVENTIONS:
Drug: 68Ga-NOTA-MAL-Cys39-exendin-4 — After 68Ga-NOTA-MAL-Cys39-exendin-4 injection, the patient drank 300-500ml of water and urinated before the PET/CT scans.

SUMMARY:
Glucagon-like peptide-1 receptor (GLP-1R) is a kind of G protein coupled receptor which regulate the insulin secretion and serves as potential target in the diagnosis of functional pancreas neuroendocrine tumor. The aim of this study was the clinical evaluation of a potential GLP-1R targeted tracer 68Ga-NOTA-MAL-Cys39-exendin-4 for the detection of insulinoma.

DETAILED DESCRIPTION:
Since GLP-1R is expressed in human β-cells and highly overexpressed in insulinomas，multiple GLP-1R-targeted radiopharmaceuticals were devoted to insulinoma localization imaging.68Ga-NOTA-MAL-Cys39-exendin-4 is an optimal probe targeting GLP-1R. A single dose of 111-185 Mega-Becquerel (MBq) 68Ga-NOTA-MAL-Cys39-exendin-4 will be injected intravenously. Visual and semiquantitative method will be used to assess the PET/CT images.The investigators will determine the use of 68Ga-NOTA-MAL-Cys39-exendin-4 PET/CT in the detection of insulinomas, and to compare its diagnostic value with conventional imaging.

ELIGIBILITY:
Inclusion Criteria:

1. The patient volunteers and signs an informed consent form.
2. age ≥18 and ≤75 years old;
3. Patients with hypoglycaemia in the presence of neuroglycopenic symptoms and documented Whipple's triad;
4. Biochemically proven endogenous hyperinsulinemic hypoglycaemia (plasma glucose concentration <3.0 mM, insulin >3 µU/ml, and C-peptide >0.6 ng/ml);
5. Conventional imaging within 3 month.

Exclusion Criteria:

1. Having a history of allergy to similar drugs, allergic constitution or suffering from allergic diseases;
2. Breast feeding;
3. Pregnancy or the wish to become pregnant within 6 months;
4. Renal function: serum creatinine > 3.0 mg/dl;
5. Any medical condition that, in the opinion of the investigator, may significantly interfere with study compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-05-05 (Actual); Primary Completion 2020-04-05 (Estimated); Study Completion 2020-05-05 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value | 1 year
  Calculation of the standardized uptake value 68Ga-NOTA-MAL-Cys39-exendin-4 in Diagnosis of Insulinoma

SECONDARY OUTCOMES:
GLP-1 receptor expression by histology compared to tracer uptake | 1 year
  Pathological detection of GLP-1 receptor expression in patients' lesions and compared to tracer uptake by PET/CT
Incidence of Adverse Events | Adverse events within 1 week after the injection and scanning of patients will be followed and assessed
  This study will utilize the CTCAE (NCI Common Terminology Criteria for Adverse Events) Version 4.0 for toxicity and Serious Adverse Event reporting

CONTACTS AND LOCATIONS:
Overall Officials: Feng Wang, Ph.D, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China